CLINICAL TRIAL: NCT02127008
Title: The Impact of Epidural Fat Resection on Postoperative Outcomes in Posterior Surgery of Lumbar Spine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin S. Yeom, Seoul National University Bundang Hospital, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EFDSC-001
Record Dates: First submitted 2014-04-28; First posted 2014-04-30 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Spinal Stenosis
Keywords: epidural fat; resection; spinal stenosis; lumbar spine
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resection of epidural fat (Experimental): During surgical procedure, epidural fat was resected fully.
  Interventions: Procedure: Resection of epidural fat
- No resection of epidural fat (Active Comparator): During surgical procedure, the epidural fat was not resected.
  Interventions: Procedure: No resection of epidural fat

INTERVENTIONS:
Procedure: Resection of epidural fat — During surgical procedure, the epidural fat with pituitary forcep and rongeur was resected.
  Arms: Resection of epidural fat
Procedure: No resection of epidural fat — During surgical procedure, the epidural fat with pituitary forcep and rongeur was not resected.
  Arms: No resection of epidural fat

SUMMARY:
Posterior lumbar epidural fat commonly had been considered a simple space-filling tissue. Anatomic studies on posterior epidural space and its contents are few, including semifluid property. In other words, there has not been studied thoroughly regarding the significance and role of posterior epidural fat in lumbar spine. In adults, epidural fat situated in the posterior triangle limited by the lamina, the ligamentum flavum, and the posterior surface of thecal sac. The fat tissue was covered by a thin membrane of connective tissue, which were free under this layer. The anterior surface of this membrane lay close to the dura mater without any attachment.

To date, the epidural fat has been resected routinely by pituitary forcep and suction drainage during posterior lumbar surgery. However, the investigators focused on the role of epidural fat, which might be associated with postoperative outcome. The investigators thought that this peculiar character, epidural fat, should be caused by certain etiologies. In general, each tissue, such as epidural fat, has its inherited features and significance, thereby the epidural fat has also specific role. However, there has not been fully studies regarding it. Thus, the investigators aimed to evaluate the impact of the posterior epidural fat on the postoperative outcomes such as pain intensity and functional outcomes by whether the epidural fat would be resected or not during posterior decompressive surgery. The investigators hypothesized that the epidural fat would be associated with postoperative pain intensitive, functional outcomes, and complications of the surgery such as failed back surgery syndrome. In this study, new device for resection of epidural fat was not utilized, but just resected with conventional devices such as pituitary forcep.

ELIGIBILITY:
Inclusion Criteria:

* patients with a lumbar spinal stenosis, which were diagnosed using lumbar spine radiographs and magnetic resonance images (MRI) that corresponded to clinical manifestations and physical examinations
* patients who underwent one-level posterior decompression
* patients aging between 20 and 80 years
* patients who volunteered for this study with written consent
* patient who were followed-up for one year or more

Exclusion Criteria:

* fractures, infection, or tumors in the lumbar spine
* patients with hemorrhagic disorders such as hemophilia and thrombocythemia
* patient with a follow-up period of less than one year
* patients who are not suitable for this study judged by the principal investigator

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2013-02; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Pain score on the VAS | Postoperative 1 month
  Pain intensity at lower back and radiating pain on the lower extremity were separately recorded at postoperative 1 month using visual analogue scale (VAS).

SECONDARY OUTCOMES:
Functional outcomes with Oswestry disability index (ODI) and SF-12 | postoperative 3 and 12 months
  Functional outcome was assessed using ODI and SF-12 at the follow-up times.
The extent of epidural fibrosis | Postoperative 1 month
  the extent of epidural fibrosis was measured with the angle of leg raise at the postoperative 1 month.
The change at postoperative enhanced MRI | 3, 12 months
  epidural inflammation and postoperative change at the posterior epidural area of the affected segment was evaluated by postoperative enhanced L-spine MRI.

CONTACTS AND LOCATIONS:
Locations (1):
- Armed Forces Yangju Hospital, Yangju, Gyounggido, South Korea